CLINICAL TRIAL: NCT04163523
Title: A Single Center, Phase I, Open-Label, Randomized, Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of a Single Dose of BGB-3111 Given Orally at 320 mg QD in Healthy Adult Subjects
Brief Title: Study to Evaluate the Effect of Food on the Pharmacokinetics of a BGB-3111 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: BGB-3111-103
Record Dates: First submitted 2019-11-05; First posted 2019-11-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
Keywords: Phase 1, pharmacokinetics safety
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Sequence 1 (Experimental): 5 Subjects received Period 1- 320 mg BGB-3111 administered after an overnight fast; Period 2- 320 mg BGB-3111 administered after High Fat/Calorie Meal; Period 3 - Day 15: 320 mg BGB-3111 administered after Low Fat/Calorie Meal
  Interventions: Drug: Zanubrutinib
- Treatment Sequence 2 (Experimental): 5 Subjects received Period 1 - Day 1: 320 mg BGB-3111 administered after High Fat/Calorie Meal; Period 2- Day 8: 320 mg BGB-3111 administered after Low Fat/Calorie Meal; Period 3- Day 15: 320 mg BGB-3111 administered after an overnight fast
  Interventions: Drug: Zanubrutinib
- Treatment Sequence 3 (Experimental): Approximately 5 Subjects receive Period 1-Day 1: 320 mg BGB-3111 administered after Low Fat/Calorie Meal; Period 2-Day 8: 320 mg BGB-3111 administered after an overnight fast; Period 3- Day 15: 320 mg BGB-3111 administered after High Fat/Calorie Meal
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib
  Other Names: BGB-3111

SUMMARY:
Phase 1 study in healthy subjects to determine the effect of food on the pharmacokinetics of BGB-3111.

DETAILED DESCRIPTION:
A randomized, crossover study to evaluate the effect of food on pharmacokinetics of BGB-3111 when administered in subjects either after a high fat/calorie meal or a low fat/calorie meal or after an overnight fast.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 to 65 years of age (inclusive)
2. Subjects must be willing and able to give written informed consent by signing an IRB-approved Informed Consent Form prior to admission to this study
3. Male subjects must agree to use a medically acceptable method of contraception from Screening until 90 days after administration of the last dose of study drug. Medically acceptable methods of contraception include the following: abstinence; a condom in addition to having the female partner use another form of contraception such as medically approved hormonal methods, diaphragm, intrauterine device or a tubal ligation. This requirement may be waived if the Principal Investigator or delegate is satisfied that the subject or partner is sterile (i.e., if female has undergone a hysterectomy, or has undergone a tubal ligation at least 3 months prior to Screening, or is postmenopausal (no menstrual period for at least 12 months prior to Screening); if male has undergone vasectomy at least 6 months prior to Screening). Male subjects agrees not to donate sperm for at least 90 days after administration of the last dose of study drug
4. Female subjects of non-childbearing potential measures, meeting at least one of the following criteria:

   1. amenorrhoeal for 12 months (menopause confirmed by Follicular Stimulating Hormone (FSH) and Luteinising Hormone (LH) levels as defined by the established reference ranges), or
   2. surgically sterile (e.g. hysterectomy, oophorectomy, tubal ligation for at least 3 months)
5. Males and females with a body mass Index (BMI) range 18-35 kg/m2 inclusive.
6. Subjects who are healthy as determined by pre-study medical history, physical examination, and 12-Lead ECG
7. Subjects who have clinical laboratory test results during the screening period that are within the reference ranges or are clinically acceptable to the Investigator
8. Subjects who test negative for HIV, HBV, and HCV by standard serologic tests must be negative at Screening
9. Subjects who test negative for drugs of abuse and alcohol tests at screening and admission
10. Subjects who are nonsmokers(ex-smokers should have quit smoking at least 6 months prior to screening)

Exclusion Criteria:

1. Subjects who have a history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders that, in the Investigator's opinion, could affect the conduct of the study or the absorption, metabolism or excretion of the study drug
2. Subjects who have a history of relevant drug hypersensitivity
3. Subjects who have a history of substance abuse, drug addiction or alcoholism
4. Subjects who consume more than 14 units of alcohol per week for women and 28 units of alcohol for men
5. A QTc at screening, check-in (all periods), and pre and post study drug dosing of greater than 450 msec for males and females
6. Subjects with the following laboratory abnormalities (at Screening and check-in of each period): a leucocyte count < 4.0x10^9/L, a neutrophil count of < 2.5x10^9, lymphocyte count < 1.2x10^9/L, Haemoglobin < 10 g/L, or transaminase levels (ALT, AST) > ULN
7. Subjects who have a significant infection, an acute infection such as influenza, coryzal symptoms, recent upper respiratory tract infection, or known inflammatory process at the time of screening and/or admission
8. Subjects who have acute gastrointestinal symptoms at the time of screening and/or admission (e.g. nausea, vomiting, diarrhea, heartburn)
9. Subjects who have used prescription drugs within 14 days of first dosing, unless agreed as nonclinically relevant by the Investigator and BeiGene (hormone replacement therapy will be permitted)
10. Subjects who have used over the counter medication excluding routine vitamins and herbal supplements (paracetamol <2 grams/day is acceptable) but including mega dose vitamin therapy and St John's Wort within 7 days of first dosing and throughout the study, unless agreed as nonclinically relevant by the Investigator and BeiGene
11. Subjects who have used any investigational drug and /or participated in any clinical trial within 2 months of first dosing
12. Subjects who have donated and/or received any blood or blood products within the previous 3 months prior to first dosing. Subjects should not donate blood while on the study and for at least 60 days after last dose of study medication
13. Subjects who have consumed food or beverage (including caffeine, alcohol, and grapefruit-containing products) known to interfere with cytochrome P450 within 48 hours prior to first study drug dose
14. Subjects who cannot communicate reliably with the investigator or are unlikely to co-operate with the requirements of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2016-07-21 (Actual); Study Completion 2016-07-21 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter: Plasma concentration of zanubrutinib as measured by area under concentration-time curve (AUC(0-24)) | up to 24 hours
Pharmacokinetic Parameter: Plasma concentration of zanubrutinib as measured by area under concentration-time curve (AUC(0-∞)) | up to 2 months
Pharmacokinetic Parameter: Peak Plasma Concentration (Cmax) of zanubrutinib | up to 2 months
Pharmacokinetic Parameter: Time to Reach Peak Plasma Concentration (Tmax) of zanubrutinib | up to 2 months
Pharmacokinetic Parameter: Half-life Period of zanubrutinib (T1/2) | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: William Novotony, MD, Study Director — Beigne
Locations (5):
- Australia (5):
  - Cancer Care Wollongong, Wollongong, New South Wales
  - Austin Health, Heidelberg, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Nucleus Network, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes